CLINICAL TRIAL: NCT00399906
Title: A Phase IIa, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Clinical Efficacy, Safety, and Pharmacokinetics of Three Different Doses of BMS-582949 Given Orally to Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Study of BMS-582949 in Patients With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM119-013
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-11

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — 4-(5-(cyclopropylcarbamoyl)-2-methylphenylamino)-5-methyl-N-propylpyrrolo(1,2-f)(1,2,4)triazine-6-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A1 (Active Comparator): 10 mg
  Interventions: Drug: BMS-582949
- A2 (Active Comparator): 30 mg
  Interventions: Drug: BMS-582949
- A3 (Active Comparator): 100 mg
  Interventions: Drug: BMS-582949
- P1 (Placebo Comparator): 10 or 100 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-582949 — Tablets, Oral, Once daily, 12 weeks
  Arms: A1; A2; A3
Drug: Placebo — Tablets, Oral, Once daily, 12 weeks
  Arms: P1

SUMMARY:
The purpose of this clinical research study is to learn if BMS-582949 alone is an effective treatment for moderate to severe psoriasis. The safety of the drug and the effectiveness of each dose will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females (not nursing or not pregnant)
* 18-75 years of age
* Diagnosis of moderate to severe psoriasis for at least six months at the time of screening
* Subjects will require wash-out of certain therapies for the treatment of psoriasis but will be allowed to continue on certain topical therapies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2007-08; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the proportion of subjects achieving an IGA score of clear or almost clear at Week 12 | at Week 12

SECONDARY OUTCOMES:
Proportion of subjects achieving a PASI-50 | at Week 12
Proportion of subjects achieving a PASI-75 | at Week 12
Proportion of subjects achieving a PASI-90 | at Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (21):
- Australia (5):
  - Local Institution, Kogarah, New South Wales
  - Local Institution, Greenslopes, Queensland
  - Local Institution, North Adelaide, South Australia
  - Local Institution, Carlton, Victoria
  - Local Institution, Malvern, Victoria
- Canada (12):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Surrey, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, Oakville, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Waterloo, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution, Québec, Quebec
  - Local Institution, Saint-Léonard, Quebec
- Mexico (4):
  - Local Institution, México, Aguascalientes
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Df, Mexico City
  - Local Institution, Monterrey, Nuevo León

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx